CLINICAL TRIAL: NCT02109978
Title: Retrospective Cohort MRC ABPI STratification and Extreme Response Mechanism in Diabetes:
Brief Title: RetroMASTER - Retrospective Cohort MRC ABPI STratification and Extreme Response Mechanism in Diabetes
Acronym: RetroMASTER
Status: Completed | Type: Observational
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: University of Exeter (Other); University of Oxford (Other); Oxford University Hospitals NHS Trust (Other); University of Dundee (Other); NHS Tayside (Other Government)
Responsible Party: Sponsor
Other Study IDs: CRF117; 12/SW/0348 (Other: Research Ethics Committee)
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Diabetes
Keywords: Diabetes; Type 2 diabetes; Diabetes therapy response; Diabetes progression
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — At Visit 1 a fasting blood sample (approximately 35 mls) will be taken for DNA extraction, and to measure for markers of the progression of diabetes or response to diabetes medication and for secondary markers that may predict response. A urine sample is also collected to measure for biomarkers.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Responders: Patients with Type 2 diabetes that have been taking a second- or third-line glucose-lowering treatment (Sulphonylurea, DPP-4 inhibitors, GLP-1R agonists, SGLT2 inhibitors, Glitazone or insulin) for at least 4 months.
- Progressors: Patients with Type 2 diabetes that progressed to requiring insulin treatment ≤10 years from diagnosis or have had no requirement for insulin treatment >10 years from diagnosis.

SUMMARY:
This study will examine extreme responders to second- and third-line Type 2 Diabetes (T2D) therapy using a retrospective approach and patients with slow or fast diabetes progression.

DETAILED DESCRIPTION:
PILOT Phase (March 2013 - Dec 2014) Patients will be recruited initially from 2 centres, plus Exeter as a pre-PILOT centre. Patients with particularly good or poor response to second- and third-line Type 2 diabetes treatments and patients progressing to insulin either particularly quickly or particularly slowly will be recruited from primary, secondary, or community settings. Fasting blood and urine samples will be collected, along with standard biomeasures and information will be collected about medical history and prescribing history.

All study documentation and sample materials will be sent out to sites from the coordinating centre. Sites will be expected to process and freeze samples and send them to the Central Laboratory managed by the Chief Inspector's site where they will be analysed for genetic factors, glycaemic markers and other markers related to drug response.

POST-PILOT Phase (Jan 2015- Oct 2017): Subject to feasibility, interim analysis and continuation of funding from Medical Research Council (MRC), this project will continue for another three years.

ELIGIBILITY:
Generic Inclusion Criteria:

* Demographics: Age 18-90 inclusive
* Ethnicity: Reflective of local demographic
* Medical History: Clinical diagnosis of Type 2 diabetes
* Mental Capacity: Capacity to Consent

Responders Cohort Inclusion Criteria:

* On Sulphonylurea, DPP-4 inhibitor, GLP-1R agonist, SGLT2 inhibitor or Glitazone for > 4 months.
* Pre-treatment HbA1c≥ 58mmol/mol (7.5%).

Progressors Cohort Inclusion Criteria:

* Type 2 diabetes (not on insulin treatment within 6 months of diagnosis)
* Either: requirement for insulin treatment ≤10 years from diagnosis (defined as insulin treatment or HbA1c ≥ 69mmol/mol (8/5%) treated with two or more non-insulin diabetes therapies) or: no requirement for insulin treatment >10 years from diagnosis (defined as not on insulin treatment AND HbA1c <69mmol/mol (8.5%).

Exclusion Criteria:

* Age less than 18 years old and greater than 90 years old
* Incapacity to consent
* Type 1 diabetes.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be identified in primary care and secondary care. The method for patient identification may differ between sites and could involve:
  GP Searches; Secondary Care Clinician Referral; Research Database Searches.
Sampling Method: Non-Probability Sample
Enrollment: 562 (Actual)
Dates: Start 2013-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Response to diabetes therapy and rate of diabetes progression | Within 9 months from date of recruitment
  The primary outcome will be to compare the clinical characteristics of the patients who show an excellent response or poor response to specific second- and third- line classes of treatment for Type 2 diabetes; and of those patients that show rapid progression of Type 2 diabetes or slow progression of Type 2 diabetes to markedly high blood glucose despite the treatment that they require.

SECONDARY OUTCOMES:
Collection of samples for analysis of potential biomarkers | within 9 months of recruitment date
  To collect a set of DNA, serum and urine samples to allow analysis of potential genetic and non-genetic biomarkers for drug response and diabetes progression.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew T Hattersley, FRCP, DM, BM, Principal Investigator — University of Exeter
Locations (3):
- United Kingdom (3):
  - University of Exeter, Exeter, Devon
  - University of Oxford, Oxford, Oxfordshire
  - University of Dundee, Dundee